CLINICAL TRIAL: NCT01729585
Title: The Effects of Massage Therapy on Quality of Life in Youth and Young Adults With Cystic Fibrosis: A Pilot Study
Brief Title: The Effects of Massage Therapy on QOL in Youth/Young Adults With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#2009-0918
Record Dates: First submitted 2012-11-15; First posted 2012-11-20 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Cystic Fibrosis; Quality of Life
Keywords: cystic fibrosis; quality of life
MeSH Terms: conditions — Cystic Fibrosis | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): control group
- Massage therapy (Active Comparator): Treatment group receives pre-determined massage therapy protocol x 5 over 10-12 weeks. massage therapy protocol includes a blend of Swedish strokes and myofascial trigger point therapy. Initially, dosing will be more frequent. Treatments will be spaced out to determine the ability of the body to maintain a more efficient musculoskeletal system, especially related to respiratory and postural efforts. Each session will end with resting hands and relaxation strokes to signal the end of the session. This protocol invites increased mobility in the musculoskeletal system. The ultimate goal is to return connective tissue (including muscles and fascia) to a more relaxed and neutral state, thus allowing expansion and ease of movement of the areas of the musculoskeletal system being worked.
  Interventions: Procedure: Massage Therapy

INTERVENTIONS:
Procedure: Massage Therapy — The Massage Therapy protocol consists of a series of 5 massages administered over 10 (+2) weeks. Length of time for each visit will be approximately 1.5 - 2 hours Typically, a series of treatments over time allows the body time to integrate tissue related changes and potentially maintain a more healthy musculoskeletal state. Based on expert opinion in the field of MT, following a series of massage treatments administered over time, one can anticipate tissue changes. By adding time between treatments, data will describe the ability of subjects to maintain changes over progressively longer periods of time. Treatment protocol will be based on the application of myofascial trigger point therapy (Timberlake, 1999) to musculoskeletal areas of the body often affected by disease progression in CF.
  Arms: Massage therapy

SUMMARY:
The purpose of this study is to describe the effects of massage therapy on quality of life (QOL) in youth and young adults (ages 8 to 21 years) with cystic fibrosis (CF).

DETAILED DESCRIPTION:
Massage therapy (MT) is defined as hands on manipulation of the soft tissue of the body with the intent to produce therapeutic, physiologic effects and to promote health and well-being (Oawriter - OAC - codes.ohio.gov, 2010; American Massage Therapy Association, 2010). Quality of life is defined as a self-description (child or adult) or parent's description of the child's perceived health and well-being based on satisfaction with physical, emotional, psychosocial and school/role functioning (Varni et al., 2002). Additional measures for this study which may influence QOL include pain, pulmonary function, ease of breathing and thoracic excursion.

Research Questions:

i. What differences in changes of QOL scores, as measured by the Peds QL 4.0 (Pediatric Quality of Life Inventory) and the CFQ-R (Cystic Fibrosis Questionnaire - Revised) are found in youth and young adults with CF between the group receiving MT and control group? What changes in QOL scores in each group are found over time? ii. What differences in changes of musculoskeletal pain, as measured by the Numeric Rating Scale for pain are found in youth and young adults with CF between the group receiving MT and the control group? What changes in pain scores in each group are found over time? iii. What differences in changes of the pulmonary function are found in youth and young adults with CF between the group receiving MT and the control group in terms of the following:

1. Forced Expiratory Volume (FEV1) and Forced Vital Capacity (FVC) scores,
2. Single breath counting score, measuring ease of breathing, and
3. Thoracic excursion as measured by the cloth tape measure technique? What changes in the above pulmonary function in each group are found over time?

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Diagnosis of CF evidenced by a prior documented positive sweat test (>60 mEq/ml by quantitative pilocarpine iontophoresis and genotype with two identified mutations consistent with CF)
* Males and females, aged 8 to 21 years at time of enrollment to obtain a broad range of symptoms related to tissue changes. (Over time, individuals with CF present with increasing symptoms with age and disease progression.)
* English speaking
* Pulmonary function clinical baseline <100% (Baseline is defined as the highest PFT during the 6 months prior to PFT at enrollment.) * This criteria was eliminated to expand eligible subjects (including PFT baseline >100).
* Clinically stable as defined by no evidence of acute upper or lower respiratory tract infections or other acute illnesses requiring use of antibiotics for at least 14 days prior to enrollment. (Pulmonary exacerbation often includes cough which may affect responses to MT.) * this criteria was omitted after study began as subjects were frequently being treated with antibiotics secondary to CF and pulmonary exacerbations.
* Approval to participate from Pulmonary Physician
* Informed consent to participate

Exclusion Criteria:

* Exposed to any investigational drug or device within 30 days of enrollment
* Any other illness at time of enrollment not a direct result of CF that the pulmonary physician determines that MT is contraindicated
* Inability to lay flat on massage table as is required for massage protocol
* Platelet count within past 12 months < 100,000. (Contraindication for deep tissue MT.) *eliminated this criteria with medical approval.
* INR International Normalized Ratio (INR) - (blood test used to monitor the effectiveness of blood thinning drugs) within past 12 months > 1.5 (Delayed clotting time is a contraindication for deep tissue MT.) * eliminated this criteria with medical approval.
* History of hepatosplenomegaly as deep tissue massage is contraindicated.
* History of lung and/or liver transplant as deep tissue MT may be contraindicated with anti-rejection drug protocol.
* Received MT within the past 30 days to eliminate the potential bias of previous response to treatment. *changed protocol to allow enrollment and wait 30 days to initiate protocol.
* Skin condition or injury that would be contraindicated for MT and would restrict ability to apply massage strokes according to protocol

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Quality of life _Peds QOL and CFQ-R | measured twice; visit 1 for baseline for treatment and control group and 10-12 weeks later following last treatment for treatment group, and same time frame for control group
  standardized measures of quality of life will be administered to subject and to parents of subjects under 18 years of age. Muscle tightness, ease of breathing, and overall relaxation 0-10 scores captured subjective QOL data.

SECONDARY OUTCOMES:
Pulmonary function | pre treatment, prior to each massage, post treatment; Time 1 = initial data collection; collect data over 10-12 weeks for treatment group. For control group, time 1 is initial data collection; time 2 is 10-12 weeks later.
  Pulmonary function test will be obtained prior to first data collection visit, using clinical pft's for treatment and control groups. Clinical pft's will also be obtained for control group 10-12 weeks following first data set. For treatment group, research pft will be obtained following last massage 10-12 weeks following initial data collection.
  Ease of breathing will be measured pre and post each massage for treatment group and at time 1 and 2 for control group.
  Thoracic excursion will be measured pre and post each massage and x2 during each massage for treatment group, and at time 1 and 2 for control group.

OTHER OUTCOMES:
Pain | at time 1, obtain baseline pain score. Collect pain score pre and post each massage and 1-2 days following each massage. control group pain scores wil be obtained following timeframe for post massage data collection
  Numeric rating scale will be used to assess pain. Pain Location and NRS Pain Score __Pre massage therapy __Post massage therapy __Follow-up phone call (date)_____
  LOCATION OF PAIN NRS (0-10) Description of Pain (circle) Reported cause Start date Identify location and describe: sharp or dull; constant or intermittent Follow Up Phone Call for Pain
  Ask: "Are you having pain?" ___No ___Yes (If yes, ask the following questions and repeat for each location:
  "Where is your pain?"
  "On a scale of 0 to 10, 0 being no pain and 10 the worst pain you have ever had, rate your pain in your (location).
  How would you describe your pain in your (location)?
  Is it sharp like a stabbing knife or dull like an ache or pressure?
  Is it constant (is it steady and does not change?) or is it intermittent (does it come and go)?
  What do you think caused you to have pain in your (location)?
  When did this pain start?"

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Zink, MSN, Principal Investigator — Cincinnati Children's Hospital, Division of Child Life and Integrative Care
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Zimmer, M., Bogenschutz, L., & Zink, K. (2008). Effect of massage therapy on pain in hospitalized pediatric cystic fibrosis patients. (abstract submitted to North American Research Conference on Complementary and Integrative Medicine, 2009).